CLINICAL TRIAL: NCT01173601
Title: A Randomized, Placebo-Controlled, Double-Blind Study of LY2216684 Fixed-Dose 12 Milligrams (mg) and 18 mg Once Daily as Adjunctive Treatment for Patients With Major Depressive Disorder Who Are Partial Responders to Selective Serotonin Reuptake Inhibitor Treatment
Brief Title: A Fixed Dose Study of Adjunctive Treatment to Antidepressant Therapy for Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11316; H9P-MC-LNBM (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — alpha-((5-fluoro-2-methoxyphenyl)methyl)-alpha-(tetrahydro-2H-pyran-4-yl)-2-morpholinemethanol; Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 12 milligrams (mg) LY2216684 + SSRI (Experimental): LY2216684: 12 milligrams (mg), administered orally, once daily (QD) for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (administered orally, QD) adjunctive to their SSRI. After the CF Phase and after randomization criteria were met, participants were randomized to the LY2216684 12-mg treatment arm (AT Phase).
  Participants who completed the AT Phase or discontinued early entered a 2-week Discontinuation (DC) Phase. Participants were randomly assigned to either abrupt DC or tapered DC over the 2-week DC Phase. Participants maintained their SSRI treatment during the DC Phase.
  Interventions: Drug: LY2216684; Drug: SSRI
- 18 milligrams (mg) LY2216684 + SSRI (Experimental): LY2216684: 12 milligrams (mg), administered orally, once daily (QD) for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (administered orally, QD) adjunctive to their SSRI. After the CF Phase and after randomization criteria were met, participants were randomized to the LY2216684 18-mg treatment arm (AT Phase).
  Participants who completed the AT Phase or discontinued early entered a 2-week Discontinuation (DC) Phase. Participants were randomly assigned to either abrupt DC or tapered DC over the 2-week DC Phase. Participants maintained their SSRI treatment during the DC Phase.
  Interventions: Drug: LY2216684; Drug: SSRI
- Placebo + SSRI (Placebo Comparator): Placebo: Tablet equivalent to LY2216684, administered orally, once daily (QD) for 11 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Prior to entering the Adjunctive Treatment (AT) Phase, participants completed a 3-week Confirmation (CF) Phase where they received placebo (administered orally, QD) adjunctive to their SSRI. After the CF Phase and after randomization criteria were met, participants were randomized to the placebo treatment arm (AT Phase).
  Participants who completed the AT Phase or discontinued early had the option to enter the Discontinuation (DC) Phase. Participants who had received placebo were assigned to the abrupt DC over the 2-week DC Phase. Participants maintained their SSRI treatment during the DC Phase.
  Interventions: Drug: Placebo; Drug: SSRI

INTERVENTIONS:
Drug: LY2216684
  Other Names: Edivoxetine
  Arms: 12 milligrams (mg) LY2216684 + SSRI; 18 milligrams (mg) LY2216684 + SSRI
Drug: Placebo
  Arms: Placebo + SSRI
Drug: SSRI — Participants should have been on their SSRI for at least 6 weeks prior and were to continue on their stable dose throughout the study.
  Other Names: Selective Serotonin Reuptake Inhibitor

SUMMARY:
The primary purpose of this study is to assess whether at least 1 dose of LY2216684 (12 milligrams [mg] or 18 mg once daily) is superior to placebo once daily in the adjunctive treatment of participants with major depressive disorder (MDD) who were identified as partial responders to an adequate course of treatment with a selective serotonin reuptake inhibitor (SSRI) during an 8-week, double-blind, acute adjunctive treatment phase.

DETAILED DESCRIPTION:
Following the Confirmation Phase, participants were randomized to adjunctive LY2216684 or adjunctive placebo if they met the following randomization criteria: had <25% improvement in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score over the past 3 weeks and a current MADRS total score ≥14. Participants who did not meet criteria received adjunctive placebo to preserve the blind.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Major Depressive Disorder (MDD)
* Women of child-bearing potential may participate but must test negative for pregnancy at the time of study entry; both women/men agree to use a reliable method of birth control
* Are taking a selective serotonin reuptake inhibitor (SSRI) approved for MDD treatment within the participant's country. The SSRI prescribed, including dose, should be consistent with labeling guidelines within the participating country.
* Have a partial response to SSRI treatment
* Meet inclusion scores on pre-defined psychiatric scales to assess diagnosis of depression, disease severity, and response to SSRI treatment
* Reliable and able to keep all scheduled appointments

Exclusion Criteria:

* Presence of another primary psychiatric illness:

  * Have had or currently have any additional ongoing Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) Axis 1 condition other than major depression within 1 year of screening
  * Have had any anxiety disorder that was considered a primary diagnosis within the past year (including panic disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, and social phobia, but excluding specific phobias)
  * Have a current or previous diagnosis of a bipolar disorder, schizophrenia, or other psychotic disorder
  * Have a history of substance abuse and/or dependence within the past 1 year (drug categories defined by DSM-IV-TR), not including caffeine and nicotine
  * Have a DSM-IV-TR Axis II disorder that, in the judgment of the investigator, would interfere with compliance with protocol
* Have any diagnosed medical condition that could be exacerbated by noradrenergic agents including unstable hypertension, unstable heart disease, tachycardia, tachyarrhythmia, narrow-angle glaucoma, urinary hesitation or retention
* Use of excluded concomitant or psychotropic medication other than SSRI
* Have initiated or discontinued hormone therapy within the previous 3 months of prior to enrollment
* History of treatment resistant depression as shown by lack of response of the current depressive episode to 2 or more adequate courses of antidepressant therapy at a clinically appropriate dose for at least 4 weeks, or in the judgment of the investigator, the participant has treatment-resistant depression
* Have a lifetime history of vagal nerve stimulation, transcranial magnetic stimulation, or psychosurgery
* Have received electroconvulsive therapy in the last year
* Enrollment in a clinical study for an investigational drug
* Serious or unstable medical condition
* History of seizure disorders
* Have initiated psychotherapy or other non-drug therapies (such as acupuncture or hypnosis) within 12 weeks prior to enrollment or any time during the study. Have no change in intensity of psychotherapy within the last 6 weeks prior to enrollment or at any time during the study.
* Participants who, in the opinion of the investigator, are judged to be at serious risk for harm to self or others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1416 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (63):
- United States (22):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Habra, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Redlands, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jamaica, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allentown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Murray, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Japan (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Latvia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daugavpils
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jelgava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Liepāja
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sigulda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strenči
- Poland (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., ?Uromin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bialystok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bydgoszcz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chełmno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gorlice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Katowice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leszno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuszyn
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yekaterinburg
- South Africa (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bellville
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cape Town
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Centurion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Cape
- Ukraine (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chernihiv District
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dnipropetrovsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kherson
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Luhansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poltava
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uzhhorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia

REFERENCES:
- [Derived] Stauffer VL, Liu P, Goldberger C, Marangell LB, Nelson C, Gorwood P, Fava M. Is the Noradrenergic Symptom Cluster a Valid Construct in Adjunctive Treatment of Major Depressive Disorder? J Clin Psychiatry. 2017 Mar;78(3):317-323. doi: 10.4088/JCP.15m09972. PMID 27685842
- [Derived] Ball SG, Ferguson MB, Martinez JM, Pangallo BA, Nery ES, Dellva MA, Sparks J, Zhang Q, Liu P, Bangs M, Goldberger C. Efficacy outcomes from 3 clinical trials of edivoxetine as adjunctive treatment for patients with major depressive disorder who are partial responders to selective serotonin reuptake inhibitor treatment. J Clin Psychiatry. 2016 May;77(5):635-42. doi: 10.4088/JCP.14m09619. PMID 27035159

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The first 3 weeks was a double-blind adjunctive placebo lead-in Confirmation Phase during which participants continued their SSRI with adjunctive placebo. If randomization criteria were met, participants were randomized to receive LY2216684 12 mg, 18 mg, or placebo. If criteria were not met, participants continued on placebo to maintain the blind.
Groups:
- Placebo + SSRI (Pre-Randomized Participants): Placebo: Administered orally, once daily for 3 weeks, adjunctive to selective serotonin reuptake inhibitor (SSRI)
- 12 mg LY2216684 + SSRI (Randomized Participants): LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a SSRI
- 18 mg LY2216684 + SSRI (Randomized Participants): LY2216684: 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI
- Placebo + SSRI (Randomized Participants): Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI
- Placebo + SSRI (Non-Randomized Participants): Placebo: Administered orally, once daily for 8 weeks
Period: Confirmation (CF) Phase, 3 Weeks
Arm/Group | Placebo + SSRI (Pre-Randomized Participants) | 12 mg LY2216684 + SSRI (Randomized Participants) | 18 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-Randomized Participants)
Started | 1416 | 0 | 0 | 0 | 0
Entered Discontinuation Phase | 21 (Participants who discontinued the CF Phase had the option to enter the DC phase.) | 0 | 0 | 0 | 0
Completed | 1328 (Participants who completed the CF Phase entered the AT Phase.) | 0 | 0 | 0 | 0
Not Completed | 88 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 23 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 15 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 6 | 0 | 0 | 0 | 0
Period: Adjunctive Treatment (AT) Phase, 8 Weeks
Arm/Group | Placebo + SSRI (Pre-Randomized Participants) | 12 mg LY2216684 + SSRI (Randomized Participants) | 18 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-Randomized Participants)
Started | 0 | 231 | 230 | 240 | 627
Entered Taper Discontinuation Phase | 0 | 100 (Participants who completed the AT Phase or discontinued early entered the taper DC Phase.) | 107 (Participants who completed the AT Phase or discontinued early entered the taper DC Phase.) | 0 | 0
Entered Abrupt Discontinuation Phase | 0 | 100 (Participants who completed the AT Phase or discontinued early entered the abrupt DC Phase.) | 108 (Participants who completed the AT Phase or discontinued early entered the abrupt DC Phase.) | 221 (Participants who completed the AT Phase or discontinued early entered the abrupt DC Phase.) | 586 (Participants who completed the AT Phase or discontinued early entered the abrupt DC Phase.)
Completed | 0 | 196 | 197 | 210 | 559
Not Completed | 0 | 35 | 33 | 30 | 68
Not completed — Adverse Event | 0 | 10 | 15 | 7 | 14
Not completed — Lack of Efficacy | 0 | 10 | 6 | 8 | 9
Not completed — Lost to Follow-up | 0 | 3 | 0 | 2 | 9
Not completed — Physician Decision | 0 | 2 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 1 | 5 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 9 | 7 | 5 | 24
Not completed — Sponsor Decision | 0 | 0 | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Participants who completed the Confirmation Phase and were randomized to adjunctive LY2216684 or adjunctive placebo or who did not meet randomization criteria and continued on placebo to maintain the blind.
Groups:
- 12 mg LY2216684 + SSRI (Randomized Participants): LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- Placebo + SSRI (Non-Randomized Participants): Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI
- Total: Total of all reporting groups
Arm/Group | 12 mg LY2216684 + SSRI (Randomized Participants) | 18 mg LY2216684 + SSRI (Randomized Participants) | Placebo + SSRI (Randomized Participants) | Placebo + SSRI (Non-Randomized Participants) | Total
Number analyzed (Participants) | 231 | 230 | 240 | 627 | 1328
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.95 (12.38) | 46.06 (12.82) | 44.38 (10.60) | 44.73 (11.89) | 44.94 (11.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145 | 149 | 155 | 451 | 900
  Male | 86 | 81 | 85 | 176 | 428
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 7 | 28 | 51
  Not Hispanic or Latino | 181 | 172 | 188 | 520 | 1061
  Unknown or Not Reported | 41 | 51 | 45 | 79 | 216
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 2
  Asian | 47 | 45 | 56 | 121 | 269
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 14 | 19 | 65 | 112
  White | 164 | 170 | 164 | 429 | 927
  More than one race | 5 | 1 | 0 | 9 | 15
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 76 | 74 | 318 | 541
  Poland | 46 | 52 | 51 | 63 | 212
  Ukraine | 33 | 29 | 29 | 36 | 127
  Russia | 6 | 6 | 6 | 15 | 33
  South Africa | 10 | 9 | 10 | 44 | 73
  Latvia | 16 | 14 | 17 | 34 | 81
  Japan | 47 | 44 | 53 | 117 | 261

OUTCOME MEASURES:

1. Primary Outcome: Change From Randomization to Week 8 in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: All randomized participants who have non-missing values at the time of randomization and at least one post-randomization value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- 12 mg LY2216684 + SSRI: LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
- 18 mg LY2216684 + SSRI: LY2216684: 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI
- Placebo + SSRI: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
units on a scale | -8.47 (0.52) | -8.70 (0.53) | -7.77 (0.51)
Statistical Analysis 1: Comparison: 12 mg LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.338, Mixed Models Analysis — In order to test the primary outcome between each LY2216684 dose and placebo while controlling the overall Type I error at 0.05, the significance level was a priori partitioned equally between the 2 LY2216684 dose-placebo comparisons at 0.025
Statistical Analysis 2: Comparison: 18 mg LY2216684 + SSRI vs Placebo + SSRI; Test type: Superiority or Other; p = 0.201, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Randomization to Week 8 in Sheehan Disability Scale (SDS) Global Functional Impairment Scale
Description: The SDS was completed by the participant and used to assess the effect of the participant's symptoms on their work (Item 1), social (Item 2), and family life (Item 3). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. The Global Function Impairment Score is the sum of the 3 items, and scores ranged from 0 to 30 with higher values indicating disruption in the participant's work life (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 222 | 236
units on a scale | -5.36 (0.44) | -5.27 (0.44) | -4.47 (0.43)

3. Secondary Outcome: Change From Randomization to Week 8 in Fatigue Associated With Depression (FAsD) Impact Subscale Score
Description: The FAsD is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The impact subscale score was derived by taking the mean of Items 7 through 13 (applicable items only). Item 12 applied only to participants with a spouse or significant other, and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 221 | 236
units on a scale | -0.74 (0.06) | -0.66 (0.06) | -0.53 (0.06)

4. Secondary Outcome: Percentage of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal 10 up to Week 8
Description: A MADRS total score of less than or equal to 10 was defined as remission criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6 for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants who meet criteria for remission by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
percentage of participants | 27.83 | 26.96 | 26.67

5. Secondary Outcome: Percentage of Participants Achieving a Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of Less Than or Equal 10 for at Least 2 Consecutive Measurements, Including the Participant's Last Measurement
Description: A MADRS total score of less than or equal to 10 for at least 2 consecutive measurements, including the participant's last measurement, was defined as remission criteria at last 2 consecutive visits. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6 for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants who meet criteria for remission at last 2 consecutive visits by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: All randomized participants with a baseline and at least one post-baseline value.
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
percentage of participants | 16.96 | 19.13 | 19.58

6. Secondary Outcome: Change From Randomization to Week 8 in Hospital and Anxiety and Depression Scale (HADS) Anxiety Subscale Score
Description: The HADS is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression subscale. Scores of 11 or more on either subscale were considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit, and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: All randomized participants with a baseline and at least one post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 239
units on a scale | -1.97 (0.22) | -2.05 (0.22) | -1.85 (0.22)

7. Secondary Outcome: Percentage of Participants Who Have a Greater Than or Equal to 50 Percent Improvement in the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Randomization up to Week 8
Description: A greater than or equal to 50 percent improvement (that is, a decrease from baseline) in the MADRS total score was defined as response criteria. The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist. Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Percentage of participants was calculated by dividing the number of participants meeting response criteria at last visit by the total number of participants analyzed, multiplied by 100%.
Time Frame: Randomization up to 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
percentage of participants | 30.43 | 34.35 | 27.08

8. Secondary Outcome: Change From Randomization to Week 8 in Hospital Anxiety and Depression Scale (HADS) Depression Subscale Score
Description: The HADS is a 14-item questionnaire with 2 subscales: anxiety and depression. Each item was rated on a 4-point scale (0-3), giving maximum scores of 21 for anxiety and depression subscale. Scores of 11 or more on either subscale were considered to be a significant 'case' of psychological morbidity, while scores of 8-10 represent 'borderline' and 0-7 represent 'normal'. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline subscale score, treatment-by-visit and baseline subscale score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 239
units on a scale | -3.19 (0.26) | -3.38 (0.27) | -2.76 (0.26)

9. Secondary Outcome: Change From Randomization to Week 8 in Montgomery-Asberg Depression Rating Scale (MADRS) Individual Items
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS had a 10-item checklist (sadness [apparent], sadness [reported], inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts). Items were rated on a scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
units on a scale
  Apparent sadness | -1.18 (0.08) | -1.04 (0.08) | -1.01 (0.08)
  Reported sadness | -1.21 (0.08) | -1.20 (0.08) | -1.00 (0.08)
  Inner tension | -0.71 (0.07) | -0.74 (0.07) | -0.65 (0.07)
  Reduced sleep | -0.97 (0.09) | -0.94 (0.09) | -0.83 (0.08)
  Reduced appetite | -0.82 (0.08) | -0.74 (0.08) | -0.75 (0.08)
  Concentration difficulties | -0.88 (0.08) | -1.01 (0.08) | -0.94 (0.08)
  Lassitude | -1.04 (0.08) | -1.12 (0.08) | -0.89 (0.08)
  Inability to feel | -1.05 (0.08) | -1.07 (0.08) | -0.90 (0.08)
  Pessimistic thoughts | -0.77 (0.07) | -0.74 (0.07) | -0.74 (0.07)
  Suicidal thoughts | -0.09 (0.03) | -0.13 (0.03) | -0.15 (0.03)

10. Secondary Outcome: Change From Randomization to Week 8 in Clinical Global Impressions of Severity (CGI-S)
Description: CGI-S measures severity of depression at the time of assessment compared with the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
units on a scale | -1.01 (0.07) | -1.08 (0.07) | -0.95 (0.07)

11. Secondary Outcome: Change From Randomization to Week 8 in Fatigue Associated With Depression (FAsD) Average Score and Experience Subscale Score
Description: The FAsD is a participant-rated scale with a total of 13 items. Six of the 13 items ask how often participants experience different aspects of fatigue with responses from 1 (never) to 5 (always). Seven of the 13 items ask how often fatigue impacts various aspects of the participant's lives with responses from 1 (not at all) to 5 (very much). The experience subscale score was derived by taking the mean of Items 1 through 6, and the average score was the mean of Items 1 through 13 (derived by taking the mean of all applicable items for each participant). Item 12 applied only to participants with a spouse or significant other, and Item 13 applied to participants who had a job or who went to school. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 221 | 236
units on a scale
  Average score | -0.69 (0.05) | -0.67 (0.05) | -0.57 (0.05)
  Experience score | -0.66 (0.06) | -0.67 (0.06) | -0.60 (0.05)

12. Secondary Outcome: Change From Randomization to Week 8 in Sheehan Disability Scale (SDS) Items
Description: The Sheehan Disability Scale (SDS) was completed by the participant and used to assess the effect of the participant's symptoms on their work (work/school impairment score), social life (social life/leisure activities impairment score), and family life (family life/home responsibilities impairment score). Each item is measured on a 0 (not at all) to 10 (extremely) point scale with higher values indicating greater disruption. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline item score, treatment-by-visit, and baseline item score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 222 | 236
units on a scale
  Work impairment score: number analyzed (Participants) | 149 | 145 | 167
  Work impairment score | -1.77 (0.19) | -1.74 (0.20) | -1.44 (0.19)
  Social life impairment score | -1.85 (0.16) | -1.81 (0.16) | -1.64 (0.16)
  Family life impairment score | -1.72 (0.16) | -1.71 (0.16) | -1.43 (0.15)

13. Secondary Outcome: Change From Randomization to Week 8 in the Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q-SF)
Description: The Q-LES-Q-SF is a self-administered 16-item questionnaire that measures degree of enjoyment and satisfaction experienced in various areas of daily life during the past week on a 5-point, Likert scale (1=very poor and 5=very good). The total raw score is the sum of items 1 to 14 and ranges from 14 to 70. The raw scores are converted to and expressed as the percentage of the maximum possible score. Higher scores indicate higher levels of enjoyment/satisfaction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of maximum possible score
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 222 | 236
percentage of maximum possible score | 10.51 (0.98) | 9.93 (0.98) | 8.47 (0.95)

14. Secondary Outcome: Change From Randomization to Week 8 in the EuroQol Questionnaire-5 Dimension (EQ-5D)
Description: The EQ-5D Visual Analog Scale is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score is self-reported using a visual analogue scale, marked on a scale of 0 to 100 with 0 representing the worst imaginable health state and 100 representing best imaginable health state. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 222 | 236
units on a scale | 12.201 (1.218) | 12.762 (1.225) | 9.756 (1.188)

15. Secondary Outcome: Percentage of Treatment Emergent (TE) Suicidal Ideation and Behaviors Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captured occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal ideation was defined as a 'yes' answer to any 1 of 5 suicidal ideation questions, which included a wish to be dead and 4 different categories of active suicidal ideation. Suicidal behavior was defined as a 'yes' answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation and behavior are defined as TE if not present at baseline. Percentage of participants was calculated by dividing the number of participants with suicide-related TE events by the total number of participants at risk, multiplied by 100%. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Randomization through 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
percentage of participants
  TE of suicidal ideation | 3.91 | 3.91 | 3.33
  TE of suicidal behavior: number analyzed (Participants) | 209 | 214 | 226
  TE of suicidal behavior | 0.00 | 0.47 | 0.44

16. Secondary Outcome: Change From Randomization to Week 8 in Arizona Sexual Experiences (ASEX) Scale
Description: The ASEX scale was used to assess sexual functioning in both males and females. The ASEX total score for the male and female version was calculated as the sum of the responses (rated from 1 [extremely] to 6 [no/never]) to the 5 items of the ASEX scale. Total scores ranged from 5 to 30 with higher scores indicating greater sexual dysfunction. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 222 | 220 | 233
units on a scale | -1.32 (0.26) | -1.27 (0.26) | -0.79 (0.25)

17. Secondary Outcome: Change From Randomization to Week 8 in Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (CPFQ)
Description: The CPFQ is a 7-item participant-rated questionnaire pertaining to a participant's cognitive and physical well-being. It assesses motivation, wakefulness, energy, focus, recall, word-finding difficulty, and mental acuity. Each item was scored on a 6-point scale ranging from 1 (greater than normal) to 6 (totally absent). Total scores ranged from 7 to 42. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline score, treatment-by-visit and baseline score-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 224 | 222 | 236
units on a scale | -4.70 (0.37) | -4.41 (0.38) | -3.79 (0.36)

18. Secondary Outcome: The Percentage of Participants Experiencing Treatment-Emergent Adverse Events as a Function of CYP2D6 Phenotype
Description: Treatment-emergent adverse events (TEAEs) were events that first occurred or worsened during the treatment phase. CYP2D6 functional phenotype was classified as poor metabolizer (PM) or non-poor metabolizer (non-PM). The percentage of participants who reported the TEAE is presented for each phenotype classification. Only TEAEs for which there was a statistically significant treatment-by-SSRI therapy interaction were included: tinnitus and influenza. A summary of serious and other non-serious adverse events regardless of causality is located in the Report of Adverse Events module.
Time Frame: Through 8 weeks
Population: All randomized patients who do not discontinue from the study for the reason 'Lost to follow-up' at the first post-baseline visit.
Measure: Number; unit: percentage of participants
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 144 | 140 | 157
percentage of participants
  Tinnitus non-PM | 0.00 | 0.00 | 1.27
  Tinnitus PM: number analyzed (Participants) | 77 | 83 | 76
  Tinnitus PM | 0.00 | 3.61 | 0.00
  Influenza non-PM | 1.39 | 0.00 | 0.64
  Influenza PM: number analyzed (Participants) | 77 | 83 | 76
  Influenza PM | 0.00 | 2.41 | 0.00

19. Secondary Outcome: Change From Randomization to Week 8 in Blood Pressure (BP)
Description: Blood pressure (BP) measurements were collected when the participant was in a sitting position. Three measurements of sitting BP collected at approximately 1-minute intervals at every visit were averaged and used as the value for the visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
millimeters of mercury (mmHg)
  Sitting systolic BP | 2.11 (0.57) | 3.18 (0.57) | 0.02 (0.55)
  Sitting diastolic BP | 3.57 (0.43) | 4.00 (0.43) | 0.66 (0.42)

20. Secondary Outcome: Change From Randomization to Week 8 in Pulse Rate
Description: Pulse measurements were collected when the participant was in a sitting position. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, investigator, visit, baseline value, treatment-by-visit and baseline value-by-visit.
Time Frame: Randomization, 8 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 12 mg LY2216684 + SSRI | 18 mg LY2216684 + SSRI | Placebo + SSRI
Number analyzed (Participants) | 230 | 230 | 240
beats per minute (bpm) | 8.66 (0.64) | 9.12 (0.64) | -1.41 (0.62)

21. Secondary Outcome: Pharmacokinetics: Plasma Concentrations of LY2216684
Description: A validated bioanalytical assay was used to determine plasma LY2216684 concentrations.
Time Frame: 1 week, 4 weeks, and 8 weeks
Population: Participants exposed to LY2216684 with evaluable plasma concentration values. Samples with concentrations below the lower quantification limit (BQL) of the assay were treated as missing values for the analysis and samples with incomplete dosing information were not included in the pharmacokinetics assessment.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2216684 + SSRI: LY2216684: fixed doses of 12 milligrams (mg) administered orally, once daily for 8 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI) or 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI
Arm/Group | LY2216684 + SSRI
Number analyzed (Participants) | 442
nanograms per milliliter (ng/mL)
  12 mg dose: number analyzed (Participants) | 427
  12 mg dose | 37.8 (20.7)
  18 mg dose: number analyzed (Participants) | 202
  18 mg dose | 55.3 (30.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 3-week double blind adjunctive placebo lead-in confirmation phase, the 8 week double-blind placebo-controlled adjunctive active treatment phase, and the 2-week discontinuation (DC) phase.
Description: During the 2-week DC phase, participants who received LY2216684 were randomly assigned to either abrupt DC or tapered DC over the 2-week period. Participants who had received placebo either during the adjunctive treatment phase or the lead-in confirmation phase remained on placebo during the 2-week DC phase.
Groups:
- Placebo + SSRI (Pre-randomized) CF Phase: Placebo: Administered orally, once daily for 3 weeks, adjunctive to a selective serotonin reuptake inhibitor (SSRI)
  Includes all enrolled participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-baseline visit during the Confirmation (CF) Phase.
- 12 mg LY2216684 + SSRI (Randomized) AT Phase: LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- 18 mg LY2216684 + SSRI (Randomized) AT Phase: LY2216684: 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Randomized) AT Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase
  Includes randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Non-randomized) AT Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes all non-randomized participants who did not discontinue for the reason 'Lost to Follow-up' at the first post-randomization visit during the Adjunctive Treatment (AT) Phase.
- Placebo + SSRI (Pre-randomized) Discontinuation Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes all enrolled participants who abruptly discontinued placebo after early withdrawal during the Confirmation (CF) Phase and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- 12 mg LY2216684 + SSRI (Abrupt Discontinuation Phase): LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a SSRI
  Includes all randomized participants who abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- 12 mg LY2216684 + SSRI (Taper Discontinuation Phase): LY2216684: 12 milligrams (mg), administered orally, once daily for 8 weeks, adjunctive to a SSRI
  Includes all randomized participants who tapered discontinuation of LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- 18 mg LY2216684 + SSRI (Abrupt Discontinuation Phase): LY2216684: 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI, during the adjunctive treatment phase
  Includes all randomized participants who abruptly discontinued LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- 18 mg LY2216684 + SSRI (Taper Discontinuation Phase): LY2216684: 12 mg, administered orally, once daily for 1 week, followed by 18 mg, administered orally, once daily for 7 weeks, adjunctive to a SSRI, during the adjunctive treatment phase
  Includes all randomized participants who tapered discontinuation of LY2216684 either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Randomized) Discontinuation Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes all randomized participants who discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
- Placebo + SSRI (Non-randomized) Discontinuation Phase: Placebo: Administered orally, once daily for 8 weeks, adjunctive to a SSRI, during the adjunctive treatment phase.
  Includes all non-randomized participants who discontinued placebo either at the end of the study or after early withdrawal from the study and who did not discontinue for the reason 'Lost to Follow-up' at the Discontinuation (DC) Phase visit.
Arm/Group | Placebo + SSRI (Pre-randomized) CF Phase | 12 mg LY2216684 + SSRI (Randomized) AT Phase | 18 mg LY2216684 + SSRI (Randomized) AT Phase | Placebo + SSRI (Randomized) AT Phase | Placebo + SSRI (Non-randomized) AT Phase | Placebo + SSRI (Pre-randomized) Discontinuation Phase | 12 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) | 12 mg LY2216684 + SSRI (Taper Discontinuation Phase) | 18 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) | 18 mg LY2216684 + SSRI (Taper Discontinuation Phase) | Placebo + SSRI (Randomized) Discontinuation Phase | Placebo + SSRI (Non-randomized) Discontinuation Phase
Serious Adverse Events (participants affected / at risk) | 2/1413 | 3/231 | 2/230 | 1/240 | 5/627 | 1/20 | 1/108 | 1/100 | 0/108 | 1/107 | 0/221 | 1/585
Other Adverse Events (participants affected / at risk) | 240/1413 | 71/231 | 73/230 | 36/240 | 100/627 | 3/20 | 17/108 | 15/100 | 18/108 | 19/107 | 39/221 | 106/585
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) CF Phase (N=1413) | 12 mg LY2216684 + SSRI (Randomized) AT Phase (N=231) | 18 mg LY2216684 + SSRI (Randomized) AT Phase (N=230) | Placebo + SSRI (Randomized) AT Phase (N=240) | Placebo + SSRI (Non-randomized) AT Phase (N=627) | Placebo + SSRI (Pre-randomized) Discontinuation Phase (N=20) | 12 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) (N=108) | 12 mg LY2216684 + SSRI (Taper Discontinuation Phase) (N=100) | 18 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) (N=108) | 18 mg LY2216684 + SSRI (Taper Discontinuation Phase) (N=107) | Placebo + SSRI (Randomized) Discontinuation Phase (N=221) | Placebo + SSRI (Non-randomized) Discontinuation Phase (N=585)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo + SSRI (Pre-randomized) CF Phase (N=1413) | 12 mg LY2216684 + SSRI (Randomized) AT Phase (N=231) | 18 mg LY2216684 + SSRI (Randomized) AT Phase (N=230) | Placebo + SSRI (Randomized) AT Phase (N=240) | Placebo + SSRI (Non-randomized) AT Phase (N=627) | Placebo + SSRI (Pre-randomized) Discontinuation Phase (N=20) | 12 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) (N=108) | 12 mg LY2216684 + SSRI (Taper Discontinuation Phase) (N=100) | 18 mg LY2216684 + SSRI (Abrupt Discontinuation Phase) (N=108) | 18 mg LY2216684 + SSRI (Taper Discontinuation Phase) (N=107) | Placebo + SSRI (Randomized) Discontinuation Phase (N=221) | Placebo + SSRI (Non-randomized) Discontinuation Phase (N=585)
Tachycardia (Cardiac disorders) | 4 (4) | 16 (16) | 23 (24) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 55 (57) | 11 (11) | 17 (21) | 1 (1) | 13 (13) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 6 (6) | 4 (4) | 19 (21)
Nasopharyngitis (Infections and infestations) | 43 (45) | 18 (18) | 10 (10) | 15 (15) | 34 (37) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 11 (11) | 10 (10)
Dizziness (Nervous system disorders) | 45 (48) | 8 (9) | 12 (13) | 5 (10) | 13 (16) | 0 (0) | 3 (3) | 5 (5) | 3 (4) | 8 (11) | 7 (9) | 34 (42)
Headache (Nervous system disorders) | 116 (136) | 22 (28) | 18 (18) | 14 (16) | 39 (47) | 3 (3) | 13 (29) | 7 (9) | 10 (14) | 10 (18) | 26 (36) | 69 (108)
Erectile dysfunction (Reproductive system and breast disorders) | 3/447 (3) | 2/86 (2) | 1/81 (1) | 0/85 (0) | 2/176 (2) | 1/6 (1) | 0/37 (0) | 0/41 (0) | 0/38 (0) | 0/37 (0) | 0/81 (0) | 0/168 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 17 (17) | 19 (20) | 16 (16) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 4 (7) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days